CLINICAL TRIAL: NCT02939742
Title: Does a Repeat Course of Antenatal Corticosteroids in Pregnant Women With Preterm Premature Rupture of Membranes Decrease Neonatal Morbidity?
Brief Title: Does a Rescue Course of Betamethasone in Pregnant Women With PPROM Decrease Neonatal Morbidity?
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low study recruitment
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-0280
Record Dates: First submitted 2016-09-23; First posted 2016-10-20 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: PPROM; Respiratory Distress Syndrome in Premature Infants
Keywords: preterm premature rupture of membranes; complications of prematurity; neonatal morbidity; respiratory distress syndrome; antenatal corticosteroids; betamethasone
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Respiratory Distress Syndrome In Premature Infants; Respiratory Distress Syndrome | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Betamethasone (Experimental): Women admitted with PPROM who will receive a second course of two betamethasone 12mg intramuscular (IM) injections given 24 hours apart.
  Interventions: Drug: Betamethasone
- Saline Placebo (Placebo Comparator): Women admitted with PPROM who will receive intramuscular saline placebo, given as two injections 24 hours apart.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Betamethasone — Betamethasone 12mg IM given every 24 hours for two doses
  Other Names: Celestone
  Arms: Betamethasone
Drug: Placebo — Sterile 0.9% normal saline solution given IM every 24 hours for two doses
  Other Names: Saline placebo
  Arms: Saline Placebo

SUMMARY:
The purpose of this study is to determine if a repeat course of betamethasone given to pregnant women with preterm premature rupture of membranes (PPROM) will decrease the infant's length of stay in the neonatal intensive care unit (NICU) and the overall neonatal morbidity associated with this condition.

DETAILED DESCRIPTION:
While the fetal benefits of a repeat course of antenatal corticosteroids have been demonstrated in several randomized controlled studies, to the investigators' knowledge they have not been adequately demonstrated in women with PPROM. Given the potential benefit of a repeat course of antenatal corticosteroids in women with PPROM on decreasing neonatal morbidity and the reassuring data from various cohorts on its safety, the investigators sought to propose a randomized controlled trial (RCT) with the hypothesis that a repeat course of antenatal corticosteroids in women with PPROM decreases neonatal morbidity.

Objectives

1. To evaluate the impact of maternal treatment with a second course of betamethasone on infant length of stay in the NICU.
2. To evaluate the impact of maternal treatment with a second course of betamethasone on the duration of neonatal need for oxygen supplementation.
3. To evaluate the impact of maternal treatment with a second course of betamethasone on neonatal morbidity overall.

Hypotheses The investigators hypothesize that treatment of women with PPROM between 24 and 34 weeks of gestation with a repeat course of antenatal corticosteroids decreases infant length of stay in the NICU and neonatal morbidity.

Aim To describe and compare the neonatal outcomes of PPROM infants exposed to a repeat course of antenatal corticosteroids compared to infants in the same antenatal conditions who are exposed to only one betamethasone course.

Subject Safety and Data Monitoring This study does not place subjects at risk of their safety. This medication is well studied and known to be safe in pregnancy.

Data monitoring will be performed and viewed by study personnel only. The data will be de-identified and a study number will be assigned to each patient. The patient's identity will be secured on a UTMB encrypted laptop device and a hard copy stored in the locked file cabinet in the locked office of the principal investigator.

Procedures to Maintain Confidentiality:

Data will be viewed by study personnel only. The data will then be de-identified and a study number will be assigned to each patient. The patient's identity will then be secured on a UTMB encrypted laptop device and a hard copy stored in the locked file cabinet in the locked office of the principal investigator.

Potential Benefits The potential benefits to subjects participating in the study include possible decreased neonatal morbidity and length of stay in the NICU.

Biostatistics Using data from the University of Texas Medical Branch (UTMB) on women with PPROM between 24 and 34 weeks, who fit the inclusion criteria, and who received the standard one course of betamethasone, the average length of stay in the NICU was 59.3 ± 36.3 days. The gestational age at delivery in this cohort was 26.5 ± 3.2 weeks.

Assuming that a second course of betamethasone reduces the length of stay needed in the NICU by 35%, and for a power of 80% and alpha 0.05, it is anticipated that enrollment of 49 women in each group will be needed, or 98 women total.

At UTMB, there are approximately 400 women per year hospitalized with PPROM. Assuming 50% of eligible women consent, the investigators estimate to finish recruitment for this study in 1-2 years.

Sample Size and Assumptions

1. Frequency of primary outcome in control group (single course of betamethasone): is 59.3 days. The investigators assume a 35% reduction in length of NICU stay using two courses of betamethasone.
2. α = 0.05, two sided
3. β = 0.2
4. Effect size: 35% reduction in primary outcome

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18 years
* Preterm premature rupture of membranes, demonstrated clinically by speculum exam
* Cervical dilation visually ≤ 5cm on sterile speculum exam
* Planned delivery at John Sealy Hospital (JSH)
* Gestational age of membrane rupture and initiation of first course of antenatal corticosteroids between 23 5/7 - 32 5/7 weeks
* Planned pregnancy continuation with no indication for delivery for at least 7 days

Exclusion Criteria:

* Maternal age > 50 years
* Gestational age < 23 5/7 weeks or > 32 5/7 weeks
* Known major congenital abnormalities, aneuploidy, or genetic syndrome
* Intrauterine fetal demise
* Any indication for expedited delivery
* Maternal chorioamnionitis
* Known allergy or adverse reaction to corticosteroids

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-11; Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Length of stay in the neonatal intensive care unit (NICU) | daily from birth of infant up to one year
  expressed in days

SECONDARY OUTCOMES:
Composite neonatal morbidity | assessed daily up to 120 days after birth or discharge from hospital, whichever occurs first
  defined as ≥ 1 of the following: RDS (oxygen requirement, clinical diagnosis, and consistent chest radiograph), bronchopulmonary dysplasia (requirement for oxygen support at 30 days of life), severe IVH (grades III or IV), periventricular leukomalacia, blood culture-proven sepsis, necrotizing enterocolitis, or perinatal death (stillbirth or death before neonatal hospital discharge)
Duration of oxygen and ventilatory support | assessed daily up to 120 days after birth or discharge from hospital, whichever occurs first
  Amount of time in days from birth that the infant requires supplemental oxygen of any form, including nasal cannula, positive airway pressure, or ventilatory support
Development of Respiratory Distress Syndrome (RDS) | assessed daily up to 120 days after birth or discharge from hospital, whichever occurs first
  Will be quantified as either present or absent. RDS defined as: compatible symptoms with radiographic evidence of hyaline membrane disease or respiratory insufficiency of prematurity requiring ventilatory support for ≥ 24 hrs
Grade III or IV intraventricular hemorrhage (IVH) | assessed daily up to 120 days after birth or discharge from hospital, whichever occurs first
  Will be quantified as either present or absent. Grade III IVH defined as ventricles enlarged by accumulating blood. Grade IV IVH defined as bleeding extending into brain matter around the ventricles.
Neonatal Sepsis | daily up to 72 hours of life
  confirmed by culture in the first 72 hours of life
Necrotizing enterocolitis (NEC) stage 2 or 3 | assessed daily up to 120 days after birth or discharge from hospital, whichever occurs first
  Will be quantified as either present or absent. Stage 2 NEC will be defined as mild to moderate systemic illness, absent bowel sounds, abdominal tenderness, pneumatosis intestinalis or portal venous gas, metabolic acidosis, decreased platelets. Stage 3 NEC will be defined as severely ill, marked distention, signs of peritonitis, hypotension, metabolic & respiratory acidosis, disseminated intravascular coagulopathy, pneumoperitoneum if bowel perforation present.
Perinatal death | assessed daily up to 120 days after birth or discharge from hospital, whichever occurs first
  defined as stillbirth or death before neonatal discharge

OTHER OUTCOMES:
Labor latency | time from admission to delivery up to one year, or through study completion
  time from diagnosis of PPROM from admission until delivery of neonate or until completion of the study
Infectious morbidities | time from admission until maternal discharge from the hospital and up until 6 weeks postpartum, or through study completion
  Chorioamnionitis will be defined as at least one temperature elevation above 38°C combined with at least two of the following signs: maternal or fetal tachycardia, uterine tenderness, foul smelling vaginal discharge, white blood count > 18,000. Postpartum endometritis will be defined as postpartum temperature elevation above 38°C without other localizing sources of infection and with either uterine tenderness or foul-smelling lochia.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bush, MD, Principal Investigator — University of Texas Medical Branch in Galveston
Locations (1):
- University of Texas Medical Branch in Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atarod Z, Taghipour M, Roohanizadeh H, Fadavi S, Taghavipour M. Effects of single course and multicourse betamethasone prior to birth in the prognosis of the preterm neonates: A randomized, double-blind placebo-control clinical trial study. J Res Med Sci. 2014 Aug;19(8):715-9. PMID 25422655
- [Background] Brookfield KF, El-Sayed YY, Chao L, Berger V, Naqvi M, Butwick AJ. Antenatal corticosteroids for preterm premature rupture of membranes: single or repeat course? Am J Perinatol. 2015 May;32(6):537-44. doi: 10.1055/s-0034-1396690. Epub 2014 Dec 29. PMID 25545441
- [Background] Elimian A, Verma U, Canterino J, Shah J, Visintainer P, Tejani N. Effectiveness of antenatal steroids in obstetric subgroups. Obstet Gynecol. 1999 Feb;93(2):174-9. doi: 10.1016/s0029-7844(98)00400-1. PMID 9932550
- [Background] Elimian A, Verma U, Visintainer P, Tejani N. Effectiveness of multidose antenatal steroids. Obstet Gynecol. 2000 Jan;95(1):34-6. doi: 10.1016/s0029-7844(99)00471-8. PMID 10636498
- [Background] Gyamfi-Bannerman C, Son M. Preterm premature rupture of membranes and the rate of neonatal sepsis after two courses of antenatal corticosteroids. Obstet Gynecol. 2014 Nov;124(5):999-1003. doi: 10.1097/AOG.0000000000000460. PMID 25437730
- [Background] Mazumder P, Dutta S, Kaur J, Narang A. Single versus multiple courses of antenatal betamethasone and neonatal outcome: a randomized controlled trial. Indian Pediatr. 2008 Aug;45(8):661-7. PMID 18723909
- [Background] National Institutes of Health Consensus Development Panel. Antenatal corticosteroids revisited: repeat courses - National Institutes of Health Consensus Development Conference Statement, August 17-18, 2000. Obstet Gynecol. 2001 Jul;98(1):144-50. doi: 10.1016/s0029-7844(01)01410-7. PMID 11430973
- [Background] Practice bulletins No. 139: premature rupture of membranes. Obstet Gynecol. 2013 Oct;122(4):918-930. doi: 10.1097/01.AOG.0000435415.21944.8f. PMID 24084566
- [Background] Wijnberger LD, Mostert JM, van Dam KI, Mol BW, Brouwers H, Visser GH. Comparison of single and repeated antenatal corticosteroid therapy to prevent neonatal death and morbidity in the preterm infant. Early Hum Dev. 2002 Apr;67(1-2):29-36. doi: 10.1016/s0378-3782(01)00248-1. PMID 11893433
- [Background] Yang SH, Choi SJ, Roh CR, Kim JH. Multiple courses of antenatal corticosteroid therapy in patients with preterm premature rupture of membranes. J Perinat Med. 2004;32(1):42-8. doi: 10.1515/JPM.2004.007. PMID 15008385